CLINICAL TRIAL: NCT00958945
Title: Retrospective & Prospective Evaluation/Analysis of Hb/Hct in Patients Having Received FloSeal (5ml &10ml) When Undergoing Total Knee or Total Hip Arthroplasty
Brief Title: Retrospective Chart Analysis in the Effective Use of FloSeal in Post-Operative Joint Replacements
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Desert Orthopedic Center Medical Research Foundation (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: John H. Velyvis, MD, Desert Orthopedic Center Medical Research Foundation
Other Study IDs: FloSeal
Record Dates: First submitted 2009-08-12; First posted 2009-08-14 (Estimated); Last update posted 2009-08-14 (Estimated); Status verified 2009-08

CONDITIONS: Total Knee Arthroplasty; Arthroplasty, Replacement, Hip
Keywords: Postoperative Hematocrit; Postoperative Hemoglobin

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- FloSeal - Knee - control: 100 Historical Control Patients, knees - no FloSeal (retrospective)
- FloSeal - Knee - 5ml: 100 Patients, knees - 5mL FloSeal (retrospective)
- FloSeal - Knee - 10ml: 100 Patients, knees- 10mL FloSeal (prospective)
- FloSeal - Hip - Control: 100 Historical Control patients, hips-no FloSeal (retrospective)
- FloSeal - Hip - 5ml: 100 retrospective patients, hips-5mL of FloSeal (retrospective)

SUMMARY:
The purpose of this analysis is to compare Hemoglobin and Hematocrit levels following total hip or knee arthroplasty. The utilization of FloSeal intraoperatively will improve hemostasis postoperatively. Decreasing bleeding time will decrease the drop in level of Hemoglobin and Hematocrit which usually occurs postoperatively.

DETAILED DESCRIPTION:
Retrospective Analysis of charts on patients having undergone Total Hip or Total Knee Arthroplasty. During the patient's hospitalization, lab values of Hg and Hct will be recorded for further analysis. Preoperative levels will be also noted to establish baselines.

Primary Data interest will be Hemoglobin (Hgb) level documented during hospitalization along with Hematocrit (HCT) and Red Blood Cell (RBC) data also collected.

Secondary Data gathered will consist of the following:

* patient Demographics
* Component Profile
* Length of Stay
* Anesthesia used
* Anesthesiologist
* EBL
* drain type
* Amount of drainage fluid recorded at 12 hour increments until discharge
* Amount of FloSeal used
* Type of Arthroplasty

  500 patients in Total
* 100 Historical Control Patients, knees - no FloSeal (retrospective)
* 100 Patients, knees - 5mL FloSeal (retrospective)
* 100 Patients, knees- 10mL FloSeal (prospective)
* 100 Historical Control patients, hips-no FloSeal (retrospective)
* 100 retrospective patients, hips-5mL of FloSeal (retrospective

Patients scheduled for Total Knee Arthroplasty will be asked if they wish to participate in the part of the study utilizing 10mL of FloSeal. These patient will be consented and the their data will be retrospectively gathered.

ELIGIBILITY:
Inclusion Criteria:

* Total Knee and Total Hip Patients
* Surgical Time less than 2 hours

Exclusion Criteria:

* Patients who require greater than 2 hour surgeries
* Patients who are undergoing revision arthroplasty
* Patients with known allergies to materials of bovine origin

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Dr. Velyvis's patients that have had a Total Knee or Total Hip after January 1, 2007
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-09

CONTACTS AND LOCATIONS:
Overall Officials: John H. Velyvis,, MD, Principal Investigator — Desert Orthopedic Center
Locations (1):
- Desert Orthopedic Center, Rancho Mirage, California, United States